CLINICAL TRIAL: NCT03545932
Title: Self-perception of Health Status and Physical Condition of Elderly People Practitioners of Hydrogymnastics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Castelo Branco (Other)
Responsible Party: Principal Investigator, Carlos Farinha, Principal Investigator, Instituto Politécnico de Castelo Branco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IPCasteloBranco
Record Dates: First submitted 2018-04-20; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Physical Disability
Keywords: Hydrogymnastics; Physical Condition; Physical Activity and Health; Gerontomotricity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydrogymnastics (Experimental): Hydrogymnastics Program
  Interventions: Other: exercise program hydrogymnastics

INTERVENTIONS:
Other: exercise program hydrogymnastics — 4 months of practice hydrogymnastics

SUMMARY:
The researcher interest in self-perception of health status and physical condition of the elderly is determinant in an increasingly aging society and where one should seek to improve their quality of life.

DETAILED DESCRIPTION:
Introduction: The researcher interest in self-perception of health status and physical condition of the elderly is determinant in an increasingly aging society and where one should seek to improve their quality of life.

Objective: To study the self-perception of health status and the impact of a physical activity program oriented during 4 months in an elderly population practitioners of hydrogymnastics.

Methods: As instruments were used the questionnaire mos short health survey - 36 items version 2 (SF-36), and the battery of Functional Tests Fitness Test. The questionnaires were filled by the elderly with the presence of the investigator and the physical fitness was evaluated following the protocol of proof. The sample was constituted of 83 elderly individuals over 55 years of age. In statistical terms we used a percentage analysis in the questionnaire and in the evaluation of the physical condition after application of the Kolmogorov-Smirnov test, we used the non-parametric test for two paired variables Wilcoxon.

ELIGIBILITY:
Inclusion Criteria:

* hydrogymnastics practitioners
* participants over 55 years of age

Exclusion Criteria:

-

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2014-11-17 (Actual); Study Completion 2015-03-20 (Actual)

PRIMARY OUTCOMES:
Self-perception of health status | 1 month
  Questionnaire SF-36

SECONDARY OUTCOMES:
Muscle strength - Legs | 1 month
  Fit up and sit in the chair
Muscle strength - Arms | 1 month
  Arm curl
Flexibility - Legs | 1 month
  Sit and reach
Flexibility - Arms | 1 month
  Reach behind the back
Dynamic balance | 1 month
  Timed up and go

IPD SHARING:
Plan to Share IPD: Undecided